CLINICAL TRIAL: NCT03008915
Title: Targeting Pulmonary Perfusion in Alpha-1 Antitrypsin Deficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Alpha-1 Foundation (Other); Stony Wold-Herbert Fund, Inc. (Other)
Responsible Party: Principal Investigator, Carrie Aaron, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: AAAP9855
Record Dates: First submitted 2016-12-22; First posted 2017-01-04 (Estimated); Results first posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-01

CONDITIONS: Alpha-1 Antitrypsin Deficiency; Emphysema; Chronic Obstructive Pulmonary Disease
Keywords: alpha-1 antitrypsin deficiency; Emphysema; chronic obstructive pulmonary disease
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Emphysema; Pulmonary Disease, Chronic Obstructive | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin first then placebo (Active Comparator): Aspirin 81mg for 2 weeks followed by a washout period and then placebo for 2 weeks
  Interventions: Drug: Aspirin; Drug: Placebo; Other: Withdrawal from alpha1 antitrypsin replacement therapy
- Placebo first then aspirin (Placebo Comparator): Placebo for 2 weeks followed by a washout period and then aspirin 81mg for 2 weeks
  Interventions: Drug: Aspirin; Drug: Placebo; Other: Withdrawal from alpha1 antitrypsin replacement therapy

INTERVENTIONS:
Drug: Aspirin — 81mg aspirin taken once per day in the morning
Drug: Placebo — placebo taken once per day in the morning
Other: Withdrawal from alpha1 antitrypsin replacement therapy — After the completion of the randomization to aspirin and placebo, participants who are on alpha1 replacement therapy are asked to withhold their usual alpha1 antitrypsin replacement therapy for 5 weeks. This is not randomized.

SUMMARY:
The aim of this study is to test whether aspirin improves endothelial function in alpha-1 antitrypsin deficiency-associated lung disease, measured by pulmonary microvascular blood flow on magnetic resonance imaging (MRI) and with apoptotic endothelial microparticles.

DETAILED DESCRIPTION:
Emphysema is a common type of lung disease in patients with alpha-1 antitrypsin deficiency (AATD). Emphysema refers to destruction of the fine network of air spaces and blood vessels in the lung, and results in what looks like "holes" in the lung. Emphysema is associated with an increased risk of death but currently no medications, except for replacement of alpha-1 antitrypsin (AAT), have been shown to treat emphysema.

The study plans to enroll subjects with alpha-1 antitrypsin deficiency-associated lung disease (PiZZ phenotype) to perform a cross-over randomized controlled trial (RCT) of aspirin compared to placebo to test the hypotheses that aspirin is effective in improving blood flow in the lungs and reducing damage to the endothelial cells. Subjects will be randomized to receive aspirin or placebo for 2 weeks. There will be a 2-week washout period, then the participant will be crossed over to receive the other treatment (those who received aspirin first will receive the placebo and those who received the placebo first will receive aspirin).

Participants who are on alpha-1 replacement therapy who have had fewer than 2 exacerbations in the last year will be asked whether they are interested in a withdrawal study. For this second part of the study, eligible and willing participants will be asked to stop their alpha-1 replacement therapy for 5 weeks and come in for a 4th study visit. This will allow AAT levels to drop briefly to those seen in the absence of AAT augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Alpha-1 antitrypsin deficiency (PiZZ genotype)
* 40 years of age or older
* Evidence of emphysema on CT scan as read by a Radiologist

Exclusion Criteria:

* Platelet count < 150,000/dL, history of intracranial hemorrhage or severe GI bleed, use of systemic anticoagulant, physician prescribed use of antiplatelet drug (including aspirin and P2Y12 receptor inhibitors), or known severe liver disease
* Immunosuppression by use of medications (including oral prednisone), or those with immunomodulatory disease (organ transplantation, autoimmune conditions or actively-treated malignancy)
* Known atrial fibrillation or left ventricular (LV) systolic heart failure
* Contraindication to MRI, including pregnancy, weight > 300 lbs (due to weight limits of the machine), those with pacemakers, aneurysm clips, cochlear implants or other implanted electronic devices, or severe claustrophobia;
* Chronic renal insufficiency (estimated GFR < 45 L/min/1.73 m2 or self report) due to slightly increased risk of nephrogenic systemic fibrosis from gadolinium administration and aspirin-related renal insufficiency
* Exacerbation of respiratory symptoms within the previous 6 weeks, such as that requiring hospitalization, oral prednisone or antibiotics to control symptoms.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Aaron, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Aspirin First, Then Placebo: Aspirin 81mg for 2 weeks followed by a washout period and then placebo for 2 weeks
  Aspirin: 81mg aspirin taken once per day in the morning
  Placebo: placebo taken once per day in the morning
  Withdrawal from alpha1 antitrypsin replacement therapy: After the completion of the randomization to aspirin and placebo, participants who are on alpha1 replacement therapy are asked to withhold their usual alpha1 antitrypsin replacement therapy for 5 weeks. This is not randomized.
- Placebo First, Then Aspirin: Placebo for 2 weeks followed by a washout period and then aspirin 81mg for 2 weeks
  Aspirin: 81mg aspirin taken once per day in the morning
  Placebo: placebo taken once per day in the morning
  Withdrawal from alpha1 antitrypsin replacement therapy: After the completion of the randomization to aspirin and placebo, participants who are on alpha1 replacement therapy are asked to withhold their usual alpha1 antitrypsin replacement therapy for 5 weeks. This is not randomized.
Period: Treatment 1
Arm/Group | Aspirin First, Then Placebo | Placebo First, Then Aspirin
Started | 8 | 7
Completed | 8 | 6
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Treatment 2
Arm/Group | Aspirin First, Then Placebo | Placebo First, Then Aspirin
Started | 8 | 6
Completed | 8 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- Overall Study: Baseline characteristics reported for all 15 participants in the crossover study.
Arm/Group | Overall Study
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Smoking status [Count of Participants; unit: Participants]
  Former smoker | 9
  Never smoker | 6
FEV1/FVC ratio [Mean (Standard Deviation); unit: percent] | 44.0 (13.0)
Percent emphysema, -950 HU [Mean (Standard Deviation); unit: percent] — Population: 1 participant withdrew before CT scan
  percent
    number analyzed (Participants) | 14
    (all) | 21.2 (9.8)

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Microvascular Blood Flow, Mean
Description: Pulmonary microvascular blood flow is measured on contrast-enhanced MRI, limited to blood flow in the 2cm periphery of the lung
Time Frame: 2 weeks
Population: Due to errors in acquisition of MRI, a number of participants had uninterpretable scans. 13 participants had MRIs interpretable for PMBF on placebo, and 7 on aspirin. Altogether, there were 6 participants with paired results from the two scans.
Measure: Mean (Standard Deviation); unit: mL blood/minute per 100mL lung
Groups:
- Aspirin: Assessment on aspirin 81mg for 2 weeks.
- Placebo: Assessment on placebo for 2 weeks.
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 6 | 6
mL blood/minute per 100mL lung | 36.9 (13.0) | 35.1 (15.4)
Statistical Analysis 1: Comparison: Aspirin vs Placebo; The null hypothesis is that there is no difference between measures on aspirin and placebo; Test type: Other — Paired t-test for participants with measures on both aspirin and placebo; p = 0.692, t-test, 2 sided

2. Secondary Outcome: Endothelial Microparticles
Description: Endothelial microparticles (EMPs) are vesicles shed from endothelial plasma membranes into the circulation in response to endothelial cell perturbation. CD31+ is a measure of apoptotic endothelial microparticles, CD62+ (P-selectin) is a measure of endothelial activation, and Annexin V/CD31+ is a more specific marker of endothelial cell apoptosis.
Time Frame: 2 weeks
Population: Due to lab closure and technician availability, only the first 3 participants had EMPs measured.
Measure: Mean (Standard Deviation); unit: EMPs/uL
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 3 | 2
EMPs/uL
  CD31+ | 749.0 (231.1) | 821.5 (3.5)
  CD62+ | 1357.3 (469.6) | 596 (287.1)
  Annexin V, CD31+ | 145.0 (62.8) | 317.0 (210.7)

3. Secondary Outcome: Endothelial Microparticles
Description: as for outcome 2
Time Frame: 5 weeks
Population: Only 2 participants had EMPs measured on placebo and 2 off AAT replacement therapy, only 1 participant had EMPs measured at both time points.
Measure: Mean (Standard Deviation); unit: EMPs/uL
Groups:
- Off Alpha-1 Replacement Therapy: Assessment after 5 weeks off alpha-1 replacement therapy
Arm/Group | Off Alpha-1 Replacement Therapy | Placebo
Number analyzed (Participants) | 2 | 2
EMPs/uL
  CD31+ | 996.0 (408.7) | 821.5 (3.5)
  CD62+ | 3681.5 (3806.4) | 596.0 (287.1)
  Annexin V, CD31+ | 146.0 (186.7) | 317.0 (210.7)

4. Secondary Outcome: Pulmonary Microvascular Blood Flow, Mean
Description: Pulmonary microvascular blood flow is measured on contrast-enhanced MRI in the peripheral 2cm of the lung.
Time Frame: 5 weeks
Population: 2 participants who completed the withdrawal phase had MRIs interpretable for PMBF on placebo and off AAT replacement therapy, data for the other 2 participants was uninterpretable for at least 1 of the 2 scans.
Measure: Mean (Standard Deviation); unit: mL blood/minute per 100mL lung
Arm/Group | Off Alpha-1 Replacement Therapy | Placebo
Number analyzed (Participants) | 2 | 13
mL blood/minute per 100mL lung | 35.5 (2.6) | 35.1 (11.0)

ADVERSE EVENTS:
Time Frame: During the course of the study, typically this was 6 weeks, but up to 11 weeks for those also withheld their alpha-1 antitrypsin replacement therapy.
Arm/Group | Aspirin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/14 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=14) | Placebo (N=15)
Syncope (Vascular disorders) | 0 (0) | 1 (1) — Patient developed syncope during spirometry/

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT03008915/Prot_SAP_000.pdf